CLINICAL TRIAL: NCT00920205
Title: Phase 1 Study of MCP-3100 in Patients With Refractory or Relapsed Cancer
Brief Title: Safety Study of MPC-3100 in Cancer Patients Who Have Failed Other Treatments
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Myrexis Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: MPC-3100-001
Record Dates: First submitted 2009-06-12; First posted 2009-06-15 (Estimated); Last update posted 2011-10-14 (Estimated); Status verified 2011-10

CONDITIONS: Cancer
Keywords: MPC-3100; HSP90 inhibitor; oral drug; cancer
MeSH Terms: conditions — Neoplasms | interventions — 1-(4-(2-(6-amino-8-((6-bromo-1,3-benzodioxol-5-yl)sulfanyl)-9H-purin-9-yl)ethyl)piperidin-1-yl)-2-hydroxypropan-1-one

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: MPC-3100 (an Hsp90 inhibitor) — oral daily dose for 21 days in a 28-day cycle

SUMMARY:
The purpose of this study is to see how safe the study drug is and to determine the best dose to use in cancer patients in the future.

The study drug is designed to reduce the activity of a protein known as "heat shock protein 90", or "Hsp90". Hsp90 is found in every cell in the human body and normally helps those cells (and the body) cope with stressful situations. In certain cancers, however, Hsp90 helps the cancer cells survive and grow. By reducing the activity of Hsp90, the study drug may slow the growth, and reduce the survival, of those cancer cells.

DETAILED DESCRIPTION:
This is a dose escalation study. As subjects participating in the study tolerate a specific dose level, the new subjects entering will be given a higher dose of the study drug.

ELIGIBILITY:
Inclusion Criteria:

* recurrent cancer refractory to available systemic therapy
* 18 years old or older
* predicted life expectancy equal or greater to 8 weeks
* at least 4 weeks post chemotherapy, immunotherapy, surgery, or radiation therapy and have recovered from treatment toxicities
* Karnofsky Performance Status equal or greater to 60 or ECOG equal or less than 2
* adequate organ function based on hematological, liver, and renal function
* LVEF greater than the lower limit of normal for the institution, as measured by MUGA or by echocardiography
* wash-out period before first dose os study drug if a protocol prohibited medication is being discontinued

Exclusion Criteria:

* pregnant or breastfeeding
* received any other anti-cancer treatment or investigational therapy within 28 days prior to Cycle 1 Day 1
* symptoms of heart failure equal or greater to Class III (by NYHA criteria)
* impaired cardiac function or clinically significant cardiac diseases
* concurrent treatment with medications that either markedly induce or inhibit CYP3A4
* concurrent treatment with medications that have a relative risk of prolonging the QT interval or inducing torsades de pointes if treatment cannot be discontinued or switched to a different medication prior to study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability (Maximum Tolerated Dose) | After each cohort is enrolled .

SECONDARY OUTCOMES:
Study Drug Pharmacokinetics | Cycle 1
Evidence of anti-tumor activity of study drug. | After each odd cycle and end of study.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Beelen, MD, Study Director — Myrexis Inc.
Locations (3):
- United States (3):
  - Nevada Cancer Institute, Las Vegas, Nevada
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas

REFERENCES:
- [Background] Bagatell R, Whitesell L. Altered Hsp90 function in cancer: a unique therapeutic opportunity. Mol Cancer Ther. 2004 Aug;3(8):1021-30. PMID 15299085
- [Background] Maloney A, Workman P. HSP90 as a new therapeutic target for cancer therapy: the story unfolds. Expert Opin Biol Ther. 2002 Jan;2(1):3-24. doi: 10.1517/14712598.2.1.3. PMID 11772336
- See also: Myriad Pharmaceuticals Inc. is a biopharmaceutical company focused on discovering, developing, and commercializing novel small molecule drugs that address severe medical conditions, including cancer and HIV infection. — http://www.myriadpharma.com